CLINICAL TRIAL: NCT02026648
Title: Outcome of Women With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 102159-E
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- cases with cervical cancer

SUMMARY:
Squamous cell carcinoma (SCC) of the cervix has showed a marked decline in developed countries over the past 40 years, however, there has also been an increase in relative and absolute incidence of adenocarcinoma and adenosquamous carcinoma (AC) of the uterine cervix over the same period.

Our understanding of the natural history and optimal management of AC is limited. It appears that AC and SCC of the cervix behave differently. They are different in epidemiology, prognostic factors, and patterns of failure after similar treatments. Available data suggest that they may also differ in their response to treatment. We postulate that new treatment strategies specifically tailored to AC should be explored.

However, there is few data about outcome of cervical cancer in Taiwan. So we propose this proposal for retrospective analysis of clinicopathological parameters and outcomes in patients of cervical cancer, especially for cervical adenocarcinoma and adenosquamous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Time interval: from 1991 to date.
* Comprehensive surgical staging, debulking procedure, radiotherapy or chemotherapy.
* All female patients with cervical cancer who underwent treatment for cervical cancer at Far Eastern Memorial Hospital.
* All the patients diagnosed as cervical cancer, especially for women with adeno- and adenosquamous carcinoma.
* To review:

  1. Clinical data: including age at diagnosis, presenting symptoms, gravidity, parity, menstrual history, body mass index, history of diabetes, hypertension, personal history of cancer and staging.
  2. Pathologic information: deep stromal invasion, lymph-vascular space invasion, lymph node involvement, parametrium invasion, vaginal cut end and tumor size.
  3. Survival data: disease-free and overall survival.
  4. Radiation report, Chemotherapy treatment, operation, discharge and admission note.

Exclusion Criteria:

* Not comprehensive staging/debulking procedure.
* Patients who died of postoperative complications within 30 days after surgery were excluded from the survival analysis.
* Female minors or disabled persons.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the cases with cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Outcome of women with cervical cancer | 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan